CLINICAL TRIAL: NCT06307353
Title: Trends of Contraception Methods in Urban Medical Center in El_Balyana
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Georgina Fector Zaghloul, resident _family medicine in Urban Medical Center in El_Balyana, Sohag University
Other Study IDs: Soh_Med_23_12_05MS
Record Dates: First submitted 2024-02-14; First posted 2024-03-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: trends of contraception methods — family planning practice will include number of women current use of family planning methods and its type planning fot ffuture pregnancy suggested duration before next pregnancy.women'ssatisfaction with family planning services atElBalyana urban Medical Center accessibility of the site suitability of waiting time

SUMMARY:
family planning is avital primary Health care intervention that saves lives of mothers and infants empowers women and support their choices regarding their health public life and additional education .In addition family planning is considered as a short term intervention to limit population growth and manage overpopulation problems.Globally the contraception prevalance rate an indicator for family planning programs continue to face challenges in developing countries.

ELIGIBILITY:
Inclusion Criteria:

- currently married woman in the child bearing period (15_49) years old attending El_Balyana urban medical Center

Exclusion Criteria:

women who are divorced or widowed or beyond age of fertility will be excluded -

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Females
Study Population: currently married woman in the child bearing period (15_49) years old attending El_Balyana urban medical Center
  Exclusion Criteria:
  women who are divorced or widowed or beyond age of fertility will be excluded -
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2026-01-10 (Actual); Primary Completion 2026-02-10 (Actual); Study Completion 2026-02-10 (Actual)

PRIMARY OUTCOMES:
number of married women in child bearing period attending the El_Balyana Medical Center using contraception methods . | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, El Balyana, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ntoimo L. Contraception in Africa: Is the global 2030 milestone attainable? Afr J Reprod Health. 2021 Jun;25(3):9-13. doi: 10.29063/ajrh2021/v25i3.1. No abstract available. PMID 37585836
- [Background] Harris ML, Coombe J, Forder PM, Lucke JC, Bateson D, Loxton D. Young Women's Complex Patterns of Contraceptive Use: Findings from an Australian Cohort Study. Perspect Sex Reprod Health. 2020 Sep;52(3):181-190. doi: 10.1363/psrh.12158. PMID 33191577
- [Background] Pimentel J, Ansari U, Omer K, Gidado Y, Baba MC, Andersson N, Cockcroft A. Factors associated with short birth interval in low- and middle-income countries: a systematic review. BMC Pregnancy Childbirth. 2020 Mar 12;20(1):156. doi: 10.1186/s12884-020-2852-z. PMID 32164598
- [Background] Mohamed NA, Abdel-Razik MS, Salem MR. Adjustment of family planning service statistics reports to support decision-making at central and governorate level, Egypt. J Egypt Public Health Assoc. 2022 Jan 20;97(1):4. doi: 10.1186/s42506-021-00098-7. PMID 35050432